CLINICAL TRIAL: NCT04733391
Title: Effects of Delayed Growth on the Quality of Life of Children Treated for a Chronic Disease and Quality of Life Study of Their Parents and Siblings
Acronym: CROQUIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-47; 2020-A00260-36 (Other: ANSM)
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of life questionnaire — Quality of life will be evaluated using the "child" version of the VSP-A questionnaire, for patients aged 8-10 years and the "adolescent" version for those aged 11-17 years.

SUMMARY:
Chronic childhood diseases have sometimes strong repercussions on the everyday life of patients and their families, because of strict daily treatment regimens, physical limitation or effects on social life for instance In children, chronic diseases can lead to poor growth, which can of itself affect the child's quality of life.

Our proposal is therefore to study the effects of short stature on the quality of life of children with chronic diseases treated in our multidisciplinary paediatrics department.

The quality of life of the patients' relatives will also be considered.

DETAILED DESCRIPTION:
Chronic childhood diseases have sometimes strong repercussions on the everyday life of patients and their families, because of strict daily treatment regimens, physical limitation or effects on social life for instance.

The importance of considering quality of life (an overarching concept covering the effects of the disease on physical, metal, emotional, social and behavioural well-being) in the treatment of patients with chronic conditions is now well established.

Quality of life studies often focus on a specific chronic condition. Studies of multiple chronic pathologies are rarer. However, factors such as the severity of the disease, its prognosis, the constraints of the daily regimen, and the visibility of the disease can have a greater impact than the type of disease itself. Studies of specific chronic diseases have identified several factors affecting quality of life such as age, sex, disease severity, medically unexplained symptoms, family cohesion, socio-economic status, perception of the disease, the adaptation strategies used by the child or their family… It would therefore be interesting to study the effects of these factors on chronic diseases in general, irrespective of disease type.

In children, chronic diseases can lead to poor growth, which can of itself affect the child's quality of life.

Our proposal is therefore to study the effects of short stature on the quality of life of children with chronic diseases treated in our multidisciplinary paediatrics department.

The quality of life of the patients' relatives will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 18 years
* Treated in the multidisciplinary paediatrics department of the Timone Hospital
* With a chronic disease (ICD10 definition: for at least 3 months in the current year with no curative treatment available)
* For at least three months
* Requiring at least two hospital consultations per year
* Able to complete the questionnaire
* Able to speak French
* Child and parental consent

Exclusion Criteria:

* Problems understanding the questionnaire (intellectual disability, low French proficiency)
* No social security coverage

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the quality of life of children treated for a chronic disease. using the VSP-A questionnaire for children aged 11 to 18 years and the VSP-Ae questionnaire for children aged between 8 and 11 years. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No